CLINICAL TRIAL: NCT01614223
Title: A Randomized Double-Blind Clinical Trial to Investigate the Use of Autologous Conditioned Plasma (ACP) for Patients With Plantar Fasciitis
Brief Title: Autologous Conditioned Plasma (ACP) for Patients With Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Dianne Bryant, Associate Professor, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FKSCM 2010 -1
Record Dates: First submitted 2012-06-04; First posted 2012-06-07 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Plantar Fasciitis
Keywords: Plantar fasciitis; Autologous Conditioned Plasma
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Adrenal Cortex Hormones; Betamethasone; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACP treatment (Active Comparator)
  Interventions: Procedure: ACP
- Corticosteroid treatment (Active Comparator)
  Interventions: Drug: Corticosteroid (celestone) injection

INTERVENTIONS:
Procedure: ACP — Within two weeks of the initial visit, the RN, will retrieve a 10-12 mL blood sample from all patients. After the sample is retrieved, the patient will be asked to lie prone on the plinth to assist with blinding. The blood sample will be retained in the Arthrex ABS-10010S Double Syringe with Syringe Cap and then separated using a soft spin centrifuge for 5 min at 1500 rpm/rcf. Three to four mL of platelet rich plasma will be pulled into a smaller syringe that is wrapped in opaque tape to conceal the contents of the syringe. The ACP is injected into the torn region of the tendon.
  Arms: ACP treatment
Drug: Corticosteroid (celestone) injection — Preparation of the blood sample is identical for patients in this group except that the blood sample will ultimately be discarded instead of injected. The syringe is blinded with opaque tape making it identical to the ACP group syringe and injected into the torn area of the tendon.
  Arms: Corticosteroid treatment

SUMMARY:
Plantar fasciitis presents clinically as pain in the inner heal, which is the result of degeneration of the plantar fascia, an arch supporting ligament of the foot. It manifests predominantly in those subjected to sustained weight bearing or repetitive pounding activities. Plantar fasciitis is the most common cause of inferior foot pain. Although most cases resolving within 6 months, traditional treatment regiments such as orthotics and physiotherapy are occasionally unsuccessful in treating this limitation leading to chronic symptoms (Neufeld & Cerrato, 2008; Rompe, 2009; Roxas, 2005).

Platelets are central players in clotting, inflammation and the wound healing response. Research has shown the potential of platelet rich plasma to accelerate wound healing in a variety of conditions including maxillo-fascial and plastic surgery, chronic wound healing and orthopaedics. Autologous Conditioned Plasma (ACP) is a novel treatment that may accelerate the healing of injured tissue. Treatment with ACP involves taking a blood sample from the patient, isolating the platelets and injecting them back into that patient at the injury site

ELIGIBILITY:
Inclusion Criteria:

* Painful inner heel pain for longer than three months
* at least six weeks since last corticosteroid injection
* four weeks since the last anaesthetic injection, iontophoresis, ultrasound and electromyostimulation
* one week since the last NSAIDs taken
* two days since the last analgesic, heat, ice, message, stretching, or modification of night splints and orthosis.
* scores greater or equal to 5 on the VAS PFPD scale
* scores greater or equal 30 on the AOFAS scale
* scores of greater or equal to 5 on the VAS PFPD scale and 30 on the AOFAS scale

Exclusion Criteria:

* tendon rupture
* neurological or vascular insufficiencies in the painful heel
* bilateral heel pain
* Paget's disease or calcaneal fat pad atrophy
* osteomyelitis, fracture of the calcaneus, ankle inflammation
* recent infection in the treatment area, history of rheumatic diseases
* collagenosis or metabolic disorders
* immunosuppressive therapy or coagulation disturbance and/or therapy, long-term treatment with corticosteroids
* previous heel surgery
* malignant disease, diabetes mellitus, severe cardiac or respiratory disease, significant abnormalities in hepatic function
* participation in another clinical study at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Midfoot Scale (AOFAS) | 6 weeks, 3, 6 and 12 months
  Inlcudes subjective and objective assessments and has demonstrated test retest reliability, validity, sensitivity to change and responsiveness for conditions of the foot and ankle. A minimally important change is considered to be at least a 5 point change with an effect size of 0.59.

SECONDARY OUTCOMES:
Plantar Fasciitis Pain/Disability Scale (PFPD | 6 weeks, 3, 6 and 12 months
SF-12 | 6 weeks, 3,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Bryant, PhD, Study Director — The University of Western Ontario
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, London, Ontario, Canada